CLINICAL TRIAL: NCT05170841
Title: Randomized, Double-blind, Placebo-controlled, Parallel Arm Group Study Evaluating Analgesic Efficacy and Safety of Dexketoprofen Trometamol and Tramadol Hydrochloride on Moderate to Severe Acute Pain in Patients With Acute Low Back Pain
Brief Title: Study Evaluating Dexketoprofen Trometamol/Tramadol Hydrochloride Analgesic Efficacy in Acute Low Back Pain
Acronym: Dante
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menarini International Operations Luxembourg SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEIN/18/DEX-LBP/001; 2019-003656-37 (EudraCT Number)
Record Dates: First submitted 2021-11-22; First posted 2021-12-28 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — dexketoprofen trometamol; Tramadol; tramadol, dexketoprofen drug combination

STUDY DESIGN:
Intervention Model Description: 2 study phases: a single-dose phase (first 8 hours) and a multiple-dose phase starting after the single-dose phase (from 8h until Day 5).In the single-dose phase the patients will receive a single dose treatment, consisting of 1 film-coated tablet and 2 capsules which must be orally administered together at the same time (Day 1). The multiple-dose phase will begin 8 hours after the first dose. The patients assigned to Dexketoprofen/Tramadol fixed combination or Tramadol 100 mg during the single-dose phase will continue to receive the same treatment during the multiple-dose phase; however, the patients assigned to receive placebo during the single-dose phase will either receive Dexketoprofen/Tramadol fixed combination or Tramadol 100 mg during the multiple-dose phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg treatment (Active Comparator): Two phase intervention. Single Dose Phase (time 0 - time 8h) and Multiple Dose phase (time 8h - Day 5) In this arm patients will receive during each phase film coated tablets (administered as one tablet)
  Interventions: Drug: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg
- Tramadol Hydrochloride 100 mg treatment (Active Comparator): Two phase intervention. Single Dose Phase (time 0 - time 8h) and Multiple Dose Phase (time 8h - Day 5) In this arm patients will receive during each phase (administered as 2 capsules of Tramadol 50 mg)
  Interventions: Drug: Tramadol Hydrochloride 100 mg
- Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg treatment (Placebo Comparator): Two phase intervention. Single dose phase (time 0 - time 8h) and Multiple Dose Phase (time 8h - Day 5).
  SINGLE DOSE PHASE: Placebo film-coated tablets matching Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg MULTIPLE DOSE PHASE: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg film coated tablets (administered as one tablet)
  Interventions: Drug: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg; Drug: Placebo
- Placebo and Tramadol Hydrochloride 100 mg (Placebo Comparator): Two phase intervention. Single Dose Phase (time 0 - time 8h) and Multiple Dose Phase (time 8h - Day 5).
  SINGLE DOSE PHASE: Placebo capsules matching active comparator (administered as 2 capsules of Tramadol 50 mg) MULTIPLE DOSE PHASE: Tramadol Hydrochloride 100 mg (administered as 2 capsules of Tramadol 50 mg)
  Interventions: Drug: Tramadol Hydrochloride 100 mg; Drug: Placebo

INTERVENTIONS:
Drug: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg — Administered as one single tablet to be taken every 8 hours
  Other Names: Skudexa
  Arms: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg treatment; Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg treatment
Drug: Tramadol Hydrochloride 100 mg — Administered as two capsules with 50 mg each to be taken every 8 hours
  Other Names: Tramadol
  Arms: Placebo and Tramadol Hydrochloride 100 mg; Tramadol Hydrochloride 100 mg treatment
Drug: Placebo — Administered as one tablet if matching Dexketoprofen Trometamol 25 mg and Tramadol Hydrochloride 75 mg or two capsules if matching Tramadol Hydrochloride 100 mg
  Arms: Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg treatment; Placebo and Tramadol Hydrochloride 100 mg

SUMMARY:
A randomized, double-blind, study to evaluate the analgesic efficacy and safety of Dexketoprofen trometamol and Tramadol hydrochloride combination versus placebo on moderate to severe acute pain in patients with acute low back pain.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, double-dummy, parallel group, placebo-controlled study encompassing 2 study phases: a single-dose phase (first 8 hours) and a multiple-dose phase starting after the single-dose phase (from 8h until day 5).

Study population will be of male or female patients aged 18 years to 65 years with acute low back pain of moderate to severe intensity, whose onset of the current acute low back pain episode is within 48 hours prior to Screening. Patients with or without radiculopathy will be included, excluding those with neurological signs, according to the Quebec Task Force classification. Patients experiencing a new episode of low back pain will be eligible only if preceded by a period of at least 2 months without any low back pain. Patients should be free from analgesic due to previously administered pain killer (immediate or slow release formulations), according to exclusion criteria.

Approximately 612 patients will be screened to achieve 510 patients randomly assigned to study treatment.

In the single-dose phase patients will receive a single-dose treatment, consisting of 1 film-coated tablet and 2 capsules which have to be orally administered together at the same time (Day 1). The multiple-dose phase will begin 8 hours after the first dose. The patients assigned to Dexketoprofen/Tramadol fixed combination or Tramadol 100 milligram (mg) during the single-dose phase will continue to receive the same treatment during the multiple-dose phase; however, the patients assigned to receive placebo during the single-dose phase will either receive Dexketoprofen/Tramadol fixed combination or Tramadol 100 mg during the multiple-dose phase.

ELIGIBILITY:
Inclusion Criteria:

1. Properly executed written informed consent.
2. Male or female patients aged 18 years to 65 years.
3. Patients with acute low back reporting pain of at least moderate intensity at Screening (NRS score ≥ 5). The onset of the current acute low back pain episode is within 48 hours prior to Screening.
4. Patients with or without radiculopathy will be included, excluding those with neurological signs, according to the Quebec Task Force classification.
5. Naïve patients to any low back pain or patients with previous history of low back pain experiencing a new episode, preceded by a period of at least 2 months without any low back pain prior to Screening.
6. Patients free from analgesic (as per exclusion criterion 14) due to previously administered pain killer (immediate or slow release formulations), according to physician's judgment.
7. Females participating in the study must be either:

   * Females of non childbearing potential, defined as any woman who had undergone surgical sterilization (documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or is more than 2 years post menopausal (defined as no menses for 12 months);
   * Females of childbearing potential (following menarche until menopause unless permanently sterile) provided that they have a negative pregnancy test at Screening and are routinely using an effective method of birth control resulting in a low failure rate (ie, combined hormonal contraception, intrauterine device, condoms in combination with a spermicidal cream, male partner sterilization (vasectomy), bilateral tubal occlusion or total sexual abstinence) during the study treatment.
8. Mentally competent and able to understand and give written informed consent prior to Screening.
9. Compliant to undergo all visits and procedures scheduled in the Study.

Exclusion Criteria:

1. Patients who are judged by the Investigator not to be suitable candidates for the study treatments and the Rescue Medication (RM) based on their medical history, physical examination, Concomitant Medication (CM) and concurrent systemic diseases.
2. Clinically significant abnormalities in the vital signs as per Investigator's judgment.
3. Patients with acute low back pain and radiation to limb with presence of neurologic signs (focal weakness, asymmetry of reflexes, sensory loss in a dermatome, or loss of bowel, bladder, or sexual function) according to Quebec Task Force Classification.
4. History of hypersensitivity to the study treatments, RM or to any other nonsteroidal anti-inflammatory drugs (NSAIDs), or opioids.
5. Known photoallergic or phototoxic reactions during treatment with ketoprofen or fibrates.
6. History of peptic ulcer, gastrointestinal disorders when taking NSAIDs, gastrointestinal bleeding, or other active bleeding.
7. History of allergy (eg, precipitate attacks of asthma, bronchospasm, acute rhinitis, or cause nasal polyps, urticaria or angioneurotic oedema) to the study treatments, RM or to any other NSAIDs, or opioids.
8. Anamnestic mild to severe renal dysfunction, mild to severe hepatic dysfunction, as per Investigator's judgment.
9. Patients with chronic dyspepsia.
10. Patients with severe heart failure [Class III and Class IV of New York Heart Association (NYHA) Classification].
11. History of hemorrhagic diathesis and other coagulation disorders.
12. History of or current epilepsy or convulsions.
13. Patients with Crohn's disease or ulcerative colitis.
14. Patients receiving monoamine oxidase (MAO) inhibitors (a minimum of 14 days of washout must elapse prior to the Screening).
15. Treatment with topical preparations/medications within 4 hours prior to Screening, anesthetics and muscle relaxants within 8 hours prior to Screening, short-acting analgesics (eg, paracetamol) within 4 hours prior to Screening, other analgesics within 5 half-lives prior to Screening or use of an opioid within the 14 days preceding Screening.
16. Treatment with high doses of salicylates (≥3 g/day), anticoagulants, thrombolytic and antiplatelet agents, heparins, corticosteroids (except inhalers and topical agents), lithium methotrexate, used at high doses of 15 mg/week or more, hydantoins (including phenytoin) and sulphonamides, antiepileptics, antipsychotics, serotonin reuptake inhibitors and tricyclic antidepressants, and analgesics within 48 hours or 5 half-lives (whichever is the longer) prior to Screening.
17. Patients using sedatives (eg, benzodiazepines) and hypnotic agents within 8 hours before Screening.
18. Any chronic or acute painful condition other than the study indication that may interfere with the assessment of the efficacy of the study treatment.
19. Any non-pharmacological interventional therapy for low back pain (physical therapy, acupuncture, massage etc.) one month before Screening.
20. Patients with litigation related to work.
21. Patients with severe dehydration (caused by vomiting, diarrhea, or insufficient fluid intake) within one month prior to Screening.
22. Severe respiratory depression according to physician's judgment.
23. Participation in other clinical studies in the previous 4 weeks.
24. History of drug or alcohol abuse. For the purpose of the study, alcohol abuse is defined as regularly intake of more than 4 units of alcohol per day (1 unit corresponds approximately to 125 ml wine, 200 ml beer, 25 ml spirit).
25. History of any illness or condition that, in the opinion of the Investigator might pose a risk to the patient or confound the efficacy and safety results of the study.
26. Pregnant and breastfeeding women: a pregnancy test will be performed on all women of childbearing potential at Screening.
27. Patients presenting any of the contraindications reported for dexketoprofen/tramadol, tramadol or paracetamol (according to the SmPC).
28. Known or suspected serious spinal pathology (eg, metastatic, inflammatory or infective diseases of the spine, cauda equine syndrome, trauma, spinal fracture).
29. Spinal surgery within the preceding 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giustino Varrassi, Professor, Principal Investigator — University of L'Aquila
Locations (1):
- University of L'Aquila, L’Aquila, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Varrassi G, Hanna M, Coaccioli S, Fabrizzi P, Baldini S, Kruljac I, Brotons C, Perrot S. Dexketoprofen Trometamol and Tramadol Hydrochloride Fixed-Dose Combination in Moderate to Severe Acute Low Back Pain: A Phase IV, Randomized, Parallel Group, Placebo, Active-Controlled Study (DANTE). Pain Ther. 2024 Aug;13(4):1007-1022. doi: 10.1007/s40122-024-00623-4. Epub 2024 Jun 26. PMID 38922520

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment (Both Phases): Two phase intervention. Single dose phase (SDP) (time 0 - time 8h) and Multiple dose phase (MDP) (time 8h - Day 5) In this arm patients will receive during each phase film coated tablets (administered as one tablet)
  Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg: Administered as one single tablet to be taken every 8 hours
- Tramadol Hydrochloride 100 mg Treatment (Both Phases): Two phase intervention. Single dose phase (SDP) (time 0 - time 8h) and Multiple dose phase (MDP) (time 8h - Day 5) In this arm patients will receive during each phase (administered as 2 capsules of Tramadol 50 mg)
  Tramadol Hydrochloride 100 mg: Administered as two capsules with 50 mg each to be taken every 8 hours
- Placebo (SDP) Then Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment (MDP): Two phase intervention. Single Dose Phase (SDP) (time 0 - time 8h) and Multiple Dose Phase (MDP) (time 8h - Day 5).
  SINGLE DOSE PHASE: Placebo film-coated tablets matching Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg MULTIPLE DOSE PHASE: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg film coated tablets (administered as one tablet)
  Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg: Administered as one single tablet to be taken every 8 hours
  Placebo: Administered as one tablet if matching Dexketoprofen Trometamol 25 mg and Tramadol Hydrochloride 75 mg or two capsules if matching Tramadol Hydrochloride 100 mg
- Placebo (Single Dose Phase) Then Tramadol Hydrochloride 100 mg (Multiple Dose Phase): Two phase intervention. Single Dose Phase (SDP) (time 0 - time 8h) and Multiple Dose Phase (MDP) (time 8h - Day 5).
  SINGLE DOSE PHASE: Placebo capsules matching active comparator (administered as 2 capsules of Tramadol 50 mg) MULTIPLE DOSE PHASE: Tramadol Hydrochloride 100 mg (administered as 2 capsules of Tramadol 50 mg)
  Tramadol Hydrochloride 100 mg: Administered as two capsules with 50 mg each to be taken every 8 hours
  Placebo: Administered as one tablet if matching Dexketoprofen Trometamol 25 mg and Tramadol Hydrochloride 75 mg or two capsules if matching Tramadol Hydrochloride 100 mg
Period: Single Dose Phase
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment (Both Phases) | Tramadol Hydrochloride 100 mg Treatment (Both Phases) | Placebo (SDP) Then Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment (MDP) | Placebo (Single Dose Phase) Then Tramadol Hydrochloride 100 mg (Multiple Dose Phase)
Started | 211 | 207 | 59 | 61
Completed | 210 | 205 | 59 | 59
Not Completed | 1 | 2 | 0 | 2
Not completed — Adverse Event | 1 | 2 | 0 | 2
Period: Multiple Dose Phase
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment (Both Phases) | Tramadol Hydrochloride 100 mg Treatment (Both Phases) | Placebo (SDP) Then Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment (MDP) | Placebo (Single Dose Phase) Then Tramadol Hydrochloride 100 mg (Multiple Dose Phase)
Started | 210 | 205 | 59 | 59
Completed | 209 | 202 | 58 | 55
Not Completed | 1 | 3 | 1 | 4
Not completed — Adverse Event | 1 | 2 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study encompassed 2 phases:
  * Single-dose phase (first 8 h) is BASELINE
  * Multiple-dose phase starting after the single-dose phase (from t8h until Day 5).
  In the single-dose phase, the patients received a single-dose treatment. In the multiple-dose phase patients assigned to DKP.TRIS / TRAM.HCl or TRAM.HCl previously continued the same treatment while patients assigned to placebo either received DKP.TRIS / TRAM.HCl or TRAM.HCl 100 mg during the multiple-dose phase.
Groups:
- Placebo Then Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment: Two phase intervention. Single dose phase (time 0 - time 8h) and Multiple dose phase (time 8h - Day 5).
  SINGLE DOSE PHASE: Placebo film-coated tablets matching Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg MULTIPLE DOSE PHASE: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg film coated tablets (administered as one tablet)
  Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg: Administered as one single tablet to be taken every 8 hours
  Placebo: Administered as one tablet if matching Dexketoprofen Trometamol 25 mg and Tramadol Hydrochloride 75 mg or two capsules if matching Tramadol Hydrochloride 100 mg
- Placebo Then Tramadol Hydrochloride 100 mg: Two phase intervention. Single dose phase (time 0 - time 8h) and Multiple dose phase (time 8h - Day 5).
  SINGLE DOSE PHASE: Placebo capsules matching active comparator (administered as 2 capsules of Tramadol 50 mg) MULTIPLE DOSE PHASE: Tramadol Hydrochloride 100 mg (administered as 2 capsules of Tramadol 50 mg)
  Tramadol Hydrochloride 100 mg: Administered as two capsules with 50 mg each to be taken every 8 hours
  Placebo: Administered as one tablet if matching Dexketoprofen Trometamol 25 mg and Tramadol Hydrochloride 75 mg or two capsules if matching Tramadol Hydrochloride 100 mg
- Total: Total of all reporting groups
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment | Placebo Then Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Placebo Then Tramadol Hydrochloride 100 mg | Total
Number analyzed (Participants) | 211 | 207 | 59 | 61 | 538
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 210 | 205 | 58 | 61 | 534
  >=65 years | 1 | 2 | 1 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 101 | 28 | 28 | 255
  Male | 113 | 106 | 31 | 33 | 283
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 211 | 207 | 58 | 61 | 537
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to First Achieve a Numeric Rating Scale-Pain Intensity Score <4 or a Pain Intensity Reduction of ≥30% From Drug Intake Till 8 Hours After the First Dose
Description: Time to first achieve a Numeric Rating Scale-Pain Intensity (NRS-PI) score of <4 or a pain intensity reduction ≥30% from drug intake till 8 hours after the first dose.
  Numeric Rate Scale-Pain Intensity is a Patients rated Pain Intensity scale using an 11-point Numeric Rate Scale (0 no pain; 10 worst pain).
Time Frame: 8 hours from first intake (referring to first 8 hours of Single Dose Phase)
Population: The modified intent-to-treat (mITT) population included the first cohort of patients randomized to the 4 treatment arms in a 4:4:1:1 ratio. Tramadol Hydrochloride 100 mg is not applicable for primary outcome measure since the primary objective was "To evaluate the analgesic efficacy of Dexketo/Tram fixed combination versus placebo in moderate to severe acute low back pain after the first dose (first 8 hours)"
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Dexketoprofen Trometamol 25 mg/ Tramadol Hydrochloride 75 mg Treatment (Both Phases): Two phase intervention. Single dose phase (SDP) (time 0 - time 8h) and Multiple dose phase (MDP) time 8h - Day 5) In this arm patients will receive during each phase film coated tablets (administered as one tablet)
  Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg: Administered as one single tablet to be taken every 8 hours
- Placebo (SDP) Then Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment (MDP): Two phase intervention. Single dose phase (time 0 - time 8h) and Multiple dose phase (time 8h - Day 5).
  SINGLE DOSE PHASE (SDP): Placebo film-coated tablets matching Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg MULTIPLE DOSE PHASE (MDP): Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg film coated tablets (administered as one tablet)
  Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg: Administered as one single tablet to be taken every 8 hours
  Placebo: Administered as one tablet if matching Dexketoprofen Trometamol 25 mg and Tramadol Hydrochloride 75 mg or two capsules if matching Tramadol Hydrochloride 100 mg
- Placebo (Single Dose Phase) Then Tramadol Hydrochloride 100 mg (Multiple Dose Phase): Two phase intervention. Single dose phase (time 0 - time 8h) and Multiple dose phase (time 8h - Day 5).
  SINGLE DOSE PHASE (SDP): Placebo capsules matching active comparator (administered as 2 capsules of Tramadol 50 mg) MULTIPLE DOSE PHASE (MDP): Tramadol Hydrochloride 100 mg (administered as 2 capsules of Tramadol 50 mg)
  Tramadol Hydrochloride 100 mg: Administered as two capsules with 50 mg each to be taken every 8 hours
  Placebo: Administered as one tablet if matching Dexketoprofen Trometamol 25 mg and Tramadol Hydrochloride 75 mg or two capsules if matching Tramadol Hydrochloride 100 mg
Arm/Group | Dexketoprofen Trometamol 25 mg/ Tramadol Hydrochloride 75 mg Treatment (Both Phases) | Placebo (SDP) Then Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment (MDP) | Placebo (Single Dose Phase) Then Tramadol Hydrochloride 100 mg (Multiple Dose Phase)
Number analyzed (Participants) | 204 | 51 | 50
score on a scale | 105 [15 to 480] | 120 [15 to 360] | 120 [15 to 360]
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/ Tramadol Hydrochloride 75 mg Treatment (Both Phases) vs Placebo (SDP) Then Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment (MDP) vs Placebo (Single Dose Phase) Then Tramadol Hydrochloride 100 mg (Multiple Dose Phase); Test type: Superiority; p = 0.566, t-test, 2 sided

2. Secondary Outcome: Total Pain Relief (TOTPAR) at 4h After the First Dose - Single Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Description: TOTPAR was calculated as the time-weighted sum of the PAR- (VRS) scores. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), percentage of maximum TOTPAR (%max TOTPAR), and percentage of patients achieving at least 50% of maximum TOTPAR were calculated at prespecified time point points in the single and the multiple-dose phases of the study. TOTPAR minimum and maximum values were 0 to 16 for Dexketoprofen/Tramadol group and 0 to 14 for Tramadol group. TOTPAR scale ranges from 0 with no upper limit.
Time Frame: From t=o to T=4 hours
Population: The modified intent-to-treat (mITT) population included the first cohort of patients randomized to the 4 treatment arms in a 4:4:1:1 ratio. This Secondary Endpoint is to evaluate the analgesic efficacy of Dexketoprofen/Tramadol fixed combination versus Tramadol 100 mg after the first 4 h intake during Single Dose Phase. Placebo arms measurement are not applicable since, as per outcome measure title above, this outcome measure was compared only between active arms
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment
Number analyzed (Participants) | 204 | 202
score on a scale | 4.6 (3.60) | 3.8 (2.84)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment; Test type: Superiority; p = 0.013, t-test, 2 sided

3. Secondary Outcome: Total Pain Relief (TOTPAR) at 6h After the First Dose - Single Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Description: TOTPAR was calculated as the time-weighted sum of the PAR-VRS scores. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), percentage of maximum TOTPAR (%max TOTPAR), and percentage of patients achieving at least 50% of maximum TOTPAR were calculated at prespecified time point points in the single and the multiple-dose phases of the study. TOTPAR minimum and maximum values were 0 to 24 for Dexketoprofen/Tramadol group and 0 to 19 for Tramadol group. TOTPAR scale ranges from 0 with no upper limit.
Time Frame: T=0 to T=6h
Population: The modified intent-to-treat (mITT) population included the first cohort of patients randomized to the 4 treatment arms in a 4:4:1:1 ratio.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment
Number analyzed (Participants) | 204 | 203
score on a scale | 7.4 (5.52) | 6.0 (4.41)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment; Test type: Superiority; p = 0.006, t-test, 2 sided

4. Secondary Outcome: Total Pain Relief (TOTPAR) at 8h After the First Dose - Single Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Description: TOTPAR was calculated as the time-weighted sum of the PAR-VRS scores. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), percentage of maximum TOTPAR (%max TOTPAR), and percentage of patients achieving at least 50% of maximum TOTPAR were calculated at prespecified time point points in the single and the multiple-dose phases of the study. TOTPAR minimum and maximum values were 0 to 31 for Dexketoprofen/Tramadol group and 0 to 26 for Tramadol group. TOTPAR scale ranges from 0 with no upper limit.
Time Frame: From T=0 to T=8h
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment
Number analyzed (Participants) | 204 | 204
score on a scale | 10.1 (7.18) | 8.5 (5.92)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment; Test type: Superiority; p = 0.013, t-test, 2 sided

5. Secondary Outcome: Total Pain Relief (TOTPAR) at 6h After the First Dose - Single Dose Phase - Dexketoprofen/Tramadol vs Placebo
Description: TOTPAR was calculated as the time-weighted sum of the PAR-VRS scores. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), percentage of maximum TOTPAR (%max TOTPAR), and percentage of patients achieving at least 50% of maximum TOTPAR were calculated at prespecified time point points in the single and the multiple-dose phases of the study. TOTPAR minimum and maximum values were 0 to 24 for Dexketoprofen/Tramadol group and 0 to 23 for Placebo group. TOTPAR scale ranges from 0 with no upper limit.
Time Frame: From T=0 to T=6h
Population: The modified intent-to-treat (mITT) population included the first cohort of patients randomized to the 4 treatment arms in a 4:4:1:1 ratio. This Secondary Endpoint is to evaluate the analgesic efficacy of Dexketoprofen/Tramadol fixed combination versus placebo after the first dose (first 6 h) in the Single Dose Phase. Tramadol 100 mg Arm measurement is not applicable since, as per outcome measure title above, this outcome measure was compared only between Dexketoprofen/Tramadol and Placebo
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: All patients receiving Placebo of Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg fixed combination or Tramadol Hydrochloride 100 mg. This Arm present combined data value for the combined Placebo arms in the Single Dose Phase
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Placebo
Number analyzed (Participants) | 204 | 101
score on a scale | 7.4 (5.52) | 6.1 (4.37)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment; Test type: Superiority; p = 0.031, t-test, 2 sided

6. Secondary Outcome: Total Pain Relief (TOTPAR) at 8h After the First Dose - Single Dose Phase - Dexketoprofen/Tramadol vs Placebo
Description: TOTPAR was calculated as the time-weighted sum of the PAR-VRS scores. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), percentage of maximum TOTPAR (%max TOTPAR), and percentage of patients achieving at least 50% of maximum TOTPAR were calculated at prespecified time point points in the single and the multiple-dose phases of the study. TOTPAR minimum and maximum values were 0 to 31 for Dexketoprofen/Tramadol group and 0 to 27 for Placebo group. TOTPAR scale ranges from 0 with no upper limit.
Time Frame: Form T=0 to T=8h
Population: The modified intent-to-treat (mITT) population included the first cohort of patients randomized to the 4 treatment arms in a 4:4:1:1 ratio.This Secondary Endpoint is to evaluate the analgesic efficacy of Dexketoprofen/Tramadol fixed combination versus placebo after the first dose (first 8 h) in the Single Dose Phase. Tramadol 100 mg Arm measurement is not applicable since, as per outcome measure title above, this outcome measure was compared only between Dexketoprofen/Tramadol and Placebo
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: All patients receiving Placebo of DexketoprofenTrometamol 25 mg/Tramadol Hydrochloride 75 mg fixed combination or Tramadol Hydrochloride 100 mg.This Arm present combined data value for the combined Placebo arms in the Single Dose Phase
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Placebo
Number analyzed (Participants) | 204 | 101
score on a scale | 10.1 (7.18) | 8.4 (5.81)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment; Test type: Superiority; p = 0.027, t-test, 2 sided

7. Secondary Outcome: Percentage of Maximum TOTPAR (%Max TOTPAR) at 4 Hours After the First Dose- Single Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Description: Max TOTPAR was calculated as the theoretical maximum time-weighted sum of the PAR values for each patient. The maximum possible TOTPAR was the value of TOTPAR that would have been obtained if the patient had a complete pain relief for that observation period. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), and percentage of maximum TOTPAR (%max TOTPAR), were calculated at prespecified time points in the single and the multiple-dose phases of the study. Percentage of maximum TOTPAR minimum and maximum values were 0 to 97 and 0 to 84 respectively for Dexketoprofen/Tramadol and Tramadol group. %max TOTPAR scale ranges from 0 to 100.
Time Frame: Form T=0 to T=4h
Population: The modified intent-to-treat (mITT) population included the first cohort of patients randomized to the 4 treatment arms in a 4:4:1:1 ratio. This Secondary Endpoint is to evaluate the analgesic efficacy of Dexketoprofen/ Tramadol fixed combination versus Tramadol 100 mg after the first dose (first 4 h) in the Single Dose Phase. Placebo arms measurement are not applicable since, as per outcome measure title above, this outcome measure was compared only between active arms
Measure: Mean (Standard Deviation); unit: percentage of score on a scale
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment
Number analyzed (Participants) | 204 | 202
percentage of score on a scale | 29.1 (22.57) | 24.1 (17.92)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment; Test type: Superiority; p = 0.011, t-test, 2 sided

8. Secondary Outcome: Percentage of Maximum TOTPAR (%Max TOTPAR) at 6 Hours After the First Dose- Single Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Description: Max TOTPAR was calculated as the theoretical maximum time-weighted sum of the PAR values for each patient. The maximum possible TOTPAR was the value of TOTPAR that would have been obtained if the patient had a complete pain relief for that observation period. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), and percentage of maximum TOTPAR (%max TOTPAR) were calculated at prespecified time point points in the single and the multiple-dose phases of the study. Percentage of maximum TOTPAR minimum and maximum values were 0 to 98 for Dexketoprofen/Tramadol group and 0 to 77 for Tramadol group. %max TOTPAR scale ranges from 0 to 100.
Time Frame: Form T=0 to T=6h
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of score on a scale
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment
Number analyzed (Participants) | 204 | 203
Percentage of score on a scale | 30.9 (23.04) | 25.5 (18.56)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment; Test type: Superiority; p = 0.007, t-test, 2 sided

9. Secondary Outcome: Percentage of Maximum TOTPAR (%Max TOTPAR) at 8 Hours After the First Dose- Single Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Description: The max TOTPAR was calculated as the theoretical maximum time-weighted sum of the PAR values for each patient. The maximum possible TOTPAR was the value of TOTPAR that would have been obtained if the patient had a complete pain relief for that observation period. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), and percentage of maximum TOTPAR (%max TOTPAR) were calculated at prespecified time point points in the single and the multiple-dose phases of the study. Percentage of maximum TOTPAR minimum and maximum values were 0 to 98 for Dexketoprofen/Tramadol group and 0 to 83 for Tramadol group. %max TOTPAR scale ranges from 0 to 100.
Time Frame: Form T=0 to T=8h
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of score on a scale
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment
Number analyzed (Participants) | 204 | 204
Percentage of score on a scale | 32.1 (22.75) | 27.1 (18.59)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment; Test type: Superiority; p = 0.013, t-test, 2 sided

10. Secondary Outcome: Percentage of Maximum TOTPAR (%Max TOTPAR) at 6 Hours After the First Dose- Single Dose Phase - Dexketoprofen/Tramadol vs Placebo
Description: The max TOTPAR was calculated as the theoretical maximum time-weighted sum of the PAR values for each patient. The maximum possible TOTPAR was the value of TOTPAR that would have been obtained if the patient had a complete pain relief for that observation period. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), and percentage of maximum TOTPAR (%max TOTPAR) were calculated at prespecified time point points in the single and the multiple-dose phases of the study. Percentage of maximum TOTPAR minimum and maximum values were 0 to 98 for Dexketoprofen/Tramadol group and 0 to 94 for Placebo group. %max TOTPAR scale ranges from 0 to 100.
Time Frame: Form T=0 to T=6h
Population: The modified intent-to-treat (mITT) population included the first cohort of patients randomized to the 4 treatment arms in a 4:4:1:1 ratio.This Secondary Endpoint is to evaluate the analgesic efficacy of Dexketoprofen/ Tramadol fixed combination versus placebo after the first dose (first 6 h) in the Single Dose Phase. Tramadol 100 mg Arm measurement is not applicable since, as per outcome measure title above, this outcome measure was compared only between Dexketoprofen/Tramadol and Placebo
Measure: Mean (Standard Deviation); unit: Percentage of score on a scale
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Placebo
Number analyzed (Participants) | 204 | 101
Percentage of score on a scale | 30.9 (23.04) | 25.5 (18.12)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment; Test type: Superiority; p = 0.029, t-test, 2 sided

11. Secondary Outcome: Percentage of Maximum TOTPAR (%Max TOTPAR) at 8 Hours After the First Dose- Single Dose Phase - Dexketoprofen/Tramadol vs Placebo
Description: The max TOTPAR was calculated as the theoretical maximum time-weighted sum of the PAR values for each patient. The maximum possible TOTPAR was the value of TOTPAR that would have been obtained if the patient had a complete pain relief for that observation period. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), and percentage of maximum TOTPAR (%max TOTPAR) were calculated at prespecified time point points in the single and the multiple-dose phases of the study. Percentage of maximum TOTPAR minimum and maximum values were 0 to 98 for Dexketoprofen/Tramadol group and 0 to 83 for Placebo group. %max TOTPAR scale ranges from 0 to 100.
Time Frame: Form T=0 to T=8h
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage score on a scale
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Placebo
Number analyzed (Participants) | 204 | 101
Percentage score on a scale | 32.1 (22.75) | 26.4 (18.03)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment; Test type: Superiority; p = 0.022, t-test, 2 sided

12. Secondary Outcome: Percentage of Patients Achieving at Least 50% of Maximum TOTPAR at 4 Hours After the First Dose - Single Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Time Frame: Form T=0 to T=4h
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment
Number analyzed (Participants) | 204 | 204
percentage of patients | 20.6 | 8.8
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment; Test type: Superiority; p < 0.001, t-test, 2 sided

13. Secondary Outcome: Percentage of Patients Achieving at Least 50% of Maximum TOTPAR at 6 Hours After the First Dose - Single Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Time Frame: Form T=0 to T=6h
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment
Number analyzed (Participants) | 204 | 204
percentage of patients | 22.5 | 9.8
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment; Test type: Superiority; p < 0.001, t-test, 2 sided

14. Secondary Outcome: Percentage of Patients Achieving at Least 50% of Maximum TOTPAR at 8 Hours After the First Dose - Single Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Time Frame: Form T=0 to T=8h
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment
Number analyzed (Participants) | 204 | 204
percentage of patients | 23.5 | 11.3
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment; Test type: Superiority; p = 0.001, t-test, 2 sided

15. Secondary Outcome: Percentage of Patients Achieving at Least 50% of Maximum TOTPAR at 4 Hours After the First Dose - Single Dose Phase - Dexketoprofen/Tramadol vs Placebo
Description: TOTPAR was calculated as the time-weighted sum of the PAR-VRS scores. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), percentage of maximum TOTPAR (%max TOTPAR), and percentage of patients achieving at least 50% of maximum TOTPAR were calculated at pre-specified time point points in the single and the multiple-dose phases of the study.
Time Frame: Form T=0 to T=4h
Population: The modified intent-to-treat (mITT) population included the first cohort of patients randomized to the 4 treatment arms in a 4:4:1:1 ratio.This Secondary Endpoint is to evaluate the analgesic efficacy of Dexketoprofen Trometamol 25 mg/ Tramadol Hydrochloride 75 mg fixed combination versus placebo after the first dose (first 6 h) in the Single Dose Phase. Tramadol Hydrochloride 100 mg Arm is not reported since data of patients in that Arm are not analyzed for this Endpoint
Measure: Number; unit: percentage of patients
Groups:
- Placebo: All patients receiving Placebo of Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg fixed combination or Tramadol Hydrochloride 100 mg.This Arm present combined data value for the combined Placebo arms in the Single Dose Phase
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Placebo
Number analyzed (Participants) | 204 | 102
percentage of patients | 20.6 | 8.8
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment; Test type: Superiority; p = 0.01, t-test, 2 sided

16. Secondary Outcome: Percentage of Patients Achieving at Least 50% of Maximum TOTPAR at 6 Hours After the First Dose - Single Dose Phase - Dexketoprofen/Tramadol vs Placebo
Description: TOTPAR was calculated as the time-weighted sum of the PAR-VRS scores. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), percentage of maximum TOTPAR (%max TOTPAR), and percentage of patients achieving at least 50% of maximum TOTPAR were calculated at pre specified time point points in the single and the multiple-dose phases of the study.
Time Frame: Form T=0 to T=6h
Population: as for outcome 15
Measure: Number; unit: percentage of patients
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Placebo
Number analyzed (Participants) | 204 | 102
percentage of patients | 22.5 | 8.8
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment; Test type: Superiority; p = 0.04, t-test, 2 sided

17. Secondary Outcome: Percentage of Patients Achieving at Least 50% of Maximum TOTPAR at 8 Hours After the First Dose - Single Dose Phase - Dexketoprofen/Tramadol vs Placebo
Description: as for outcome 16
Time Frame: Form T=0 to T=8h
Population: as for outcome 15
Measure: Number; unit: percentage of patients
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Placebo
Number analyzed (Participants) | 204 | 102
percentage of patients | 23.5 | 11.8
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment; Test type: Superiority; p = 0.016, t-test, 2 sided

18. Secondary Outcome: Total Pain Relief (TOTPAR) at 24h After the First Dose - Multiple Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Description: TOTPAR was calculated as the time-weighted sum of the PAR-VRS scores. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), percentage of maximum TOTPAR (%max TOTPAR), and percentage of patients achieving at least 50% of maximum TOTPAR were calculated at prespecified time point points in the single and the multiple-dose phases of the study. TOTPAR minimum and maximum values were 0 to 96 for Dexketoprofen/Tramadol group and 0 to 90 for Tramadol group. TOTPAR scale ranges from 0 with no upper limit.
Time Frame: Form T=0 to T=24h
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment: Two phase intervention. Single dose phase (time 0 - time 8h) and Multiple dose phase (time 8h - Day 5).
  SINGLE DOSE PHASE: Placebo film-coated tablets matching Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg MULTIPLE DOSE PHASE: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg film coated tablets (administered as one tablet)
  Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg: Administered as one single tablet to be taken every 8 hours
  Placebo: Administered as one tablet if matching Dexketoprofen Trometamol 25 mg and Tramadol Hydrochloride 75 mg or two capsules if matching Tramadol Hydrochloride 100 mg
- Placebo and Tramadol Hydrochloride 100 mg: Two phase intervention. Single dose phase (time 0 - time 8h) and Multiple dose phase (time 8h - Day 5).
  SINGLE DOSE PHASE: Placebo capsules matching active comparator (administered as 2 capsules of Tramadol 50 mg) MULTIPLE DOSE PHASE: Tramadol Hydrochloride 100 mg (administered as 2 capsules of Tramadol 50 mg)
  Tramadol Hydrochloride 100 mg: Administered as two capsules with 50 mg each to be taken every 8 hours
  Placebo: Administered as one tablet if matching Dexketoprofen Trometamol 25 mg and Tramadol Hydrochloride 75 mg or two capsules if matching Tramadol Hydrochloride 100 mg
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment | Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Placebo and Tramadol Hydrochloride 100 mg
Number analyzed (Participants) | 201 | 202 | 43 | 48
score on a scale | 44.6 (20.20) | 40.9 (19.85) | 44.6 (20.2) | 40.9 (19.85)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment vs Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Placebo and Tramadol Hydrochloride 100 mg; Test type: Superiority; p = 0.045, t-test, 2 sided

19. Secondary Outcome: Total Pain Relief (TOTPAR) at 48h After the First Dose - Multiple Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Description: TOTPAR was calculated as the time-weighted sum of the PAR-VRS scores. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), percentage of maximum TOTPAR (%max TOTPAR), and percentage of patients achieving at least 50% of maximum TOTPAR were calculated at prespecified time point points in the single and the multiple-dose phases of the study. TOTPAR minimum and maximum values were 0 to 192 for Dexketoprofen/Tramadol group and 0 to 184 for Tramadol group. TOTPAR scale ranges from 0 with no upper limit.
Time Frame: Form T=0 to T=48h
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment | Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Placebo and Tramadol Hydrochloride 100 mg
Number analyzed (Participants) | 201 | 202 | 47 | 49
score on a scale | 97.8 (41.69) | 90.0 (41.88) | 97.8 (41.69) | 90.0 (41.88)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment vs Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Placebo and Tramadol Hydrochloride 100 mg; Test type: Superiority; p = 0.042, t-test, 2 sided

20. Secondary Outcome: Total Pain Relief (TOTPAR) at 72h After the First Dose - Multiple Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Description: TOTPAR was calculated as the time-weighted sum of the PAR-VRS scores. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), percentage of maximum TOTPAR (%max TOTPAR), and percentage of patients achieving at least 50% of maximum TOTPAR were calculated at prespecified time point points in the single and the multiple-dose phases of the study. TOTPAR minimum and maximum values were 0 to 288 for Dexketoprofen/Tramadol group and 0 to 280 for Tramadol group. TOTPAR scale ranges from 0 with no upper limit.
Time Frame: Form T=0 to T=72h
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment | Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Placebo and Tramadol Hydrochloride 100 mg
Number analyzed (Participants) | 201 | 202 | 47 | 49
score on a scale | 156.9 (63.83) | 144.7 (64.14) | 156.9 (63.83) | 144.7 (64.14)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment vs Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Placebo and Tramadol Hydrochloride 100 mg; Test type: Superiority; p = 0.037, t-test, 2 sided

21. Secondary Outcome: Percentage of Maximum TOTPAR (%Max TOTPAR) at 24 Hours After the First Dose- Multiple Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Description: The max TOTPAR was calculated as the theoretical maximum time-weighted sum of the PAR values for each patient. The maximum possible TOTPAR was the value of TOTPAR that would have been obtained if the patient had a complete pain relief for that observation period. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), and percentage of maximum TOTPAR (%max TOTPAR) were calculated at prespecified time point points in the single and the multiple-dose phases of the study. Percentage of maximum TOTPAR minimum and maximum values were 0 to 100 for Dexketoprofen/Tramadol group and 0 to 94 for Tramadol group. %max TOTPAR scale ranges from 0 to 100.
Time Frame: Form T=0 to T=24h
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of score on a scale
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment | Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Placebo and Tramadol Hydrochloride 100 mg
Number analyzed (Participants) | 201 | 202 | 43 | 48
Percentage of score on a scale | 46.6 (21.07) | 42.7 (20.66) | 46.6 (21.07) | 42.7 (20.66)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment vs Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Placebo and Tramadol Hydrochloride 100 mg; Test type: Superiority; p = 0.045, t-test, 2 sided

22. Secondary Outcome: Percentage of Maximum TOTPAR (%Max TOTPAR) at 48 Hours After the First Dose- Multiple Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Description: The max TOTPAR was calculated as the theoretical maximum time-weighted sum of the PAR values for each patient. The maximum possible TOTPAR was the value of TOTPAR that would have been obtained if the patient had a complete pain relief for that observation period. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), and percentage of maximum TOTPAR (%max TOTPAR) were calculated at prespecified time point points in the single and the multiple-dose phases of the study. Percentage of maximum TOTPAR minimum and maximum values were 0 to 100 for Dexketoprofen/Tramadol group and 0 to 96 for Tramadol group. %max TOTPAR scale ranges from 0 to 100.
Time Frame: Form T=0 to T=48h
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of score on a scale
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment | Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Placebo and Tramadol Hydrochloride 100 mg
Number analyzed (Participants) | 201 | 202 | 47 | 49
Percentage of score on a scale | 51.2 (21.69) | 46.9 (21.79) | 51.2 (21.69) | 46.9 (21.79)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment vs Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Placebo and Tramadol Hydrochloride 100 mg; Test type: Superiority; p = 0.029, t-test, 2 sided

23. Secondary Outcome: Percentage of Maximum TOTPAR (%Max TOTPAR) at 72 Hours After the First Dose- Multiple Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Description: The max TOTPAR was calculated as the theoretical maximum time-weighted sum of the PAR values for each patient. The maximum possible TOTPAR was the value of TOTPAR that would have been obtained if the patient had a complete pain relief for that observation period. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), and percentage of maximum TOTPAR (%max TOTPAR) were calculated at prespecified time point points in the single and the multiple-dose phases of the study. Percentage of maximum TOTPAR minimum and maximum values were 0 to 100 for Dexketoprofen/Tramadol group and 0 to 97 for Tramadol group. %max TOTPAR scale ranges from 0 to 100.
Time Frame: Form T=0 to T=72h
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of score on a scale
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment | Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Placebo and Tramadol Hydrochloride 100 mg
Number analyzed (Participants) | 201 | 202 | 47 | 49
Percentage of score on a scale | 54.7 (22.15) | 50.3 (22.24) | 54.7 (22.15) | 50.3 (22.24)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment vs Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Placebo and Tramadol Hydrochloride 100 mg; Test type: Superiority; p = 0.027, t-test, 2 sided

24. Secondary Outcome: Percentage of Maximum TOTPAR (%Max TOTPAR) at 96 Hours After the First Dose- Multiple Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Description: The max TOTPAR was calculated as the theoretical maximum time-weighted sum of the PAR values for each patient. The maximum possible TOTPAR was the value of TOTPAR that would have been obtained if the patient had a complete pain relief for that observation period. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some (meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR), and percentage of maximum TOTPAR (%max TOTPAR) were calculated at prespecified time point points in the single and the multiple-dose phases of the study. Percentage of maximum TOTPAR minimum and maximum values were 0 to 100 for Dexketoprofen/Tramadol group and 0 to 98 for Tramadol group. %max TOTPAR scale ranges from 0 to 100.
Time Frame: Form T=0 to T=96h
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of score on a scale
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment | Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Placebo and Tramadol Hydrochloride 100 mg
Number analyzed (Participants) | 201 | 202 | 48 | 49
Percentage of score on a scale | 57.7 (22.7) | 53.3 (22.82) | 57.7 (22.7) | 53.3 (22.82)
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment vs Placebo and Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Placebo and Tramadol Hydrochloride 100 mg; Test type: Superiority; p = 0.035, t-test, 2 sided

25. Secondary Outcome: Percentage of Patients Achieving at Least 50% of Maximum TOTPAR at 48 Hours After the First Dose - Multiple Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Description: as for outcome 15
Time Frame: Form T=0 to T=48h
Population: Per-protocol (PP) population included all patients in the ITT having major protocol violations that could affect the primary efficacy analysis. Protocol violations which had a major distorting influence on the primary endpoints resulted in patients being excluded from the PP population. Protocol Deviations identified during the the study conduct, as authorized in the final Protocol Deviation log, were taken into consideration in the final assignment of patients to the analysis sets.
Measure: Number; unit: Percentage of patients
Groups:
- Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment: All patients receiving DexketoprofenTrometamol 25 mg/Tramadol Hydrochloride 75 mg fixed combination. This arm present combined data value from DexketoprofenTrometamol 25 mg/Tramadol Hydrochloride 75 mg arm and from Placebo then Dexketoprofen Trometamol 25mg/Tramadol Hydrochloride 75 mg arm.
- Tramadol Hydrochloride 100 mg Treatment: All patients receiving Tramadol Hydrochloride 100 mg. This arm present combined data value from Tramadol Hydrochloride 100 mg arm and from Placebo then Tramadol Hydrochloride 100 mg arm.
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment
Number analyzed (Participants) | 235 | 230
Percentage of patients | 60 | 46.5
Statistical Analysis 1: Comparison: Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment vs Tramadol Hydrochloride 100 mg Treatment; Test type: Superiority; p = 0.001, t-test, 2 sided

26. Secondary Outcome: Percentage of Patients Achieving at Least 50% of Maximum TOTPAR at 72 Hours After the First Dose - Multiple Dose Phase - Dexketoprofen/Tramadol vs Tramadol
Description: The max TOTPAR was calculated as the theoretical maximum time-weighted sum of the PAR values for each patient. The maximum possible TOTPAR was the value of TOTPAR that would have been obtained if the patient had a complete pain relief for that observation period. The Verbal Rating Scale (VRS) is a 5-point scale to assess the pain relief. The patients were asked to answer the question 'How do you rate your pain relief?' where 0 = 'no relief', 1 = 'a little (perceptible) relief', 2 = 'some(meaningful) relief', 3 = 'lot of relief', 4 = 'complete relief'. Based on VRS, pain relief (PAR) scores, total pain relief (TOTPAR),percentage of maximum TOTPAR (%max TOTPAR), and percentage of patients achieving at least 50% of maximum TOTPAR were calculated at pre specified time point points in the single and the multiple-dose phases of the study.
Time Frame: Form T=0 to T=72h
Population: as for outcome 25
Measure: Number; unit: Percentage of patients
Groups:
- Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment: All patients receiving Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg fixed combination. This arm present combined data value from Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg arm and from Placebo then Dexketoprofen Trometamol 25mg/Tramadol Hydrochloride 75 mg arm.
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment | Tramadol Hydrochloride 100 mg Treatment
Number analyzed (Participants) | 147 | 123
Percentage of patients | 62.6 | 53.5

ADVERSE EVENTS:
Time Frame: Adverse events were collected starting from informed consent signature till the end of the study at Visit 2 (Day 6+2 Days). For the purpose of the study, in accordance to study Protocol, the AEs have been divided by study phases (i.e Single Dose Phase and Multiple Dose Phase)
Description: If a patient reports the same Adverse Event (AE) more than once within that System Organ Class/Preferred Term, then that patient will be counted only once for that System Organ Class or Preferred Term
Groups:
- Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment - MULTIPLE DOSE PHASE: Multiple dose phase (time 8h - Day 5)
  In this arm patients will receive during this phase film coated tablets (administered as one tablet):
  Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg: Administered as one single tablet to be taken every 8 hours
- Tramadol Hydrochloride 100 mg Treatment - MULTIPLE DOSE PHASE: Multiple dose phase (time 8h - Day 5)
  In this arm patients will receive during this phase (administered as 2 capsules of Tramadol 50 mg):
  Tramadol Hydrochloride 100 mg: Administered as two capsules with 50 mg each to be taken every 8 hours
- Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment - SINGLE DOSE PHASE: Single dose phase (time 0 - time 8h)
  In this arm patients will receive during this phase film coated tablets (administered as one tablet):
  Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg: Administered as one single tablet to be taken every 8 hours
- Tramadol Hydrochloride 100 mg Treatment - SINGLE DOSE PHASE: Single dose phase (time 0 - time 8h)
  In this arm patients will receive during this phase (administered as 2 capsules of Tramadol 50 mg):
  Tramadol Hydrochloride 100 mg: Administered as two capsules with 50 mg each to be taken every 8 hours
- Placebo - SINGLE DOSE PHASE: Single dose phase (time 0 - time 8h) Placebo administered as one film-coated tablets if matching Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg treatment or 2 capsules if matching Tramadol Hydrochloride 100 mg Treatment (as 2 capsules of Tramadol 50 mg).
Arm/Group | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment - MULTIPLE DOSE PHASE | Tramadol Hydrochloride 100 mg Treatment - MULTIPLE DOSE PHASE | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment - SINGLE DOSE PHASE | Tramadol Hydrochloride 100 mg Treatment - SINGLE DOSE PHASE | Placebo - SINGLE DOSE PHASE
All-Cause Mortality (participants affected / at risk) | 0/270 | 0/268 | 0/211 | 0/207 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/270 | 1/268 | 1/211 | 0/207 | 0/119
Other Adverse Events (participants affected / at risk) | 68/270 | 73/268 | 28/211 | 31/207 | 11/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment - MULTIPLE DOSE PHASE (N=270) | Tramadol Hydrochloride 100 mg Treatment - MULTIPLE DOSE PHASE (N=268) | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment - SINGLE DOSE PHASE (N=211) | Tramadol Hydrochloride 100 mg Treatment - SINGLE DOSE PHASE (N=207) | Placebo - SINGLE DOSE PHASE (N=119)
Calculus Urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment - MULTIPLE DOSE PHASE (N=270) | Tramadol Hydrochloride 100 mg Treatment - MULTIPLE DOSE PHASE (N=268) | Dexketoprofen Trometamol 25 mg/Tramadol Hydrochloride 75 mg Treatment - SINGLE DOSE PHASE (N=211) | Tramadol Hydrochloride 100 mg Treatment - SINGLE DOSE PHASE (N=207) | Placebo - SINGLE DOSE PHASE (N=119)
Nausea (Gastrointestinal disorders) | 18 (18) | 25 (25) | 8 (8) | 6 (6) | 5 (5)
Vomiting (Gastrointestinal disorders) | 13 (15) | 22 (23) | 3 (3) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 17 (17) | 16 (16) | 12 (12) | 12 (12) | 2 (2)
Somnolence (Nervous system disorders) | 12 (12) | 7 (7) | 2 (2) | 7 (7) | 2 (2)
Headache (Nervous system disorders) | 8 (9) | 5 (5) | 1 (1) | 2 (2) | 2 (2)
Asthenia (General disorders) | 5 (5) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 4 (4) | 1 (1) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
No Limitations and Caveats

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/41/NCT05170841/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT05170841/SAP_001.pdf